CLINICAL TRIAL: NCT03700333
Title: Clinical Research of S-1 Versus Pemetrexed in the Maintenance Treatment of Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: Clinical Research of S-1 Versus Pemetrexed in the Maintenance Treatment of Advanced NSNSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NHP-18-01
Record Dates: First submitted 2018-09-09; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; S-1; Pemetrexed; maintenance therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-1 Group (Experimental): Stage IIIB or IV non-small-cell lung cancer (NSCLC) population treated by Tegafur,Gimeracil and Oteracil Potassium Capsules (S-1)
  Interventions: Drug: S-1 therapy
- Pemetrexed Group (Active Comparator): Stage IIIB or IV non-small-cell lung cancer (NSCLC) population treated by Pemetrexed
  Interventions: Drug: Pemetrexed therapy

INTERVENTIONS:
Drug: S-1 therapy — accept S-1(50mg, twice a day, morning and night, if<1.5m2; 75mg, twice a day, morning and night,if >1.5m2 )chemotherapy after finishing first-line therapy(>21 days).
  Arms: S-1 Group
Drug: Pemetrexed therapy — accept Pemetrexed (500mg/m2,d1)chemotherapy after finishing first-line therapy(>21 days).
  Arms: Pemetrexed Group

SUMMARY:
The purpose of this study is to compare the curative effect of oral S-1 with Pemetrexed in the maintenance treatment of advanced non-squamous non-small cell lung cancer (NSCLC), and initial to explore a new treatment strategy for advanced non-squamous NSCLC.

DETAILED DESCRIPTION:
S-1 consists of Tegafur,Gimeracil and Oteracil Potassium. Tegafur is metabolize to Gimeracil，and slows down the metabolism of 5-FU in high DPD enzyme expression tumor cell, so that 5-FU could bring the antimetabolic fiction more efficiently. Plenty of studies support that S-1 shows a desirable effect on advanced non-squamous NSCLC, and S-1 is more convenient compare with Pemetrexed. The curative effect of Pemetrexed in the maintenance treatment of advanced non-squamous NSCLC has been proved to be valid. The purpose of our study is to explore whether S-1 could replace Pemetrexed in the maintenance treatment of advanced non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histological or cytological documented
3. NSCLC of stage IIIB (surgery is unacceptable) or IV confirmed by mediastinoscopy or PET based on RECIST1.1.
4. Candidates have been accepted 4-6 cycles of gemcitabine/carboplatin Naive chemotherapy, and evaluated as CR,PR or SD.
5. Candidates's expected survival time should be greater than or equal to 3 months with ECOG performance status 0-1, adequate haematological and Hepatic- renal function, and cardiac function.
6. At least one measurable tumor lesion (maximum diameter has to be greater than 10mm scan by CT or MRI) or malignant lymph node (15mm in short axis), and must not be accepted radiotherapy.
7. No any other following malignancy or any serious complication caused by metastatic encephaloma.
8. No any gastrointestinal diseases that could reduce the drug absorption.
9. Female: Candidates who have any chance to be pregnant must accept pregnancy tests 72 hours before therapy, and take medical allowed contraceptives during therapy or in 3 mouths after therapy. Pregnancy tests results must be negative.Lactation female are not included.
10. Male: Be sterilized or take contraceptives during therapy or in 3 mouths after therapy.

Exclusion Criteria:

1. Any unstable systemic disease
2. Patients with exposure to any recent anticancer therapy outside of this trial.
3. Pregnant or breast-feeding women

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
progress free survival | 1 year
  From date of randomization until the date of first documented progression.

SECONDARY OUTCOMES:
overall survival | 3 mouths, 6 mouths, 9 mouths, 1 year
  every subjects needs to be recorded the data of death.From date of randomization until the date of death from any cause.
objective response rate | 3 mouths, 6 mouths, 9 mouths, 1 year
  ORR(objective response rate) is equal to the sum of cases of CR (complete response) and PR (partial response) divided by the total number of evaluable cases.From date of randomization until the date of first documented progression.
duration of response | 6 weeks, 3 mouths, 18 weeks, 6 mouths, 9 mouths, 1 year
  From the date of first documented CR (complete response) or PR (partial response) until the date of first documented progression or recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Shu, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University; Renhua Guo, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shirasaka T. Development history and concept of an oral anticancer agent S-1 (TS-1): its clinical usefulness and future vistas. Jpn J Clin Oncol. 2009 Jan;39(1):2-15. doi: 10.1093/jjco/hyn127. Epub 2008 Dec 3. PMID 19052037
- [Result] Kubota K, Sakai H, Yamamoto N, Kunitoh H, Nakagawa K, Takeda K, Ichinose Y, Saijo N, Ariyoshi Y, Fukuoka M. A multi-institution phase I/II trial of triweekly regimen with S-1 plus cisplatin in patients with advanced non-small cell lung cancer. J Thorac Oncol. 2010 May;5(5):702-6. doi: 10.1097/JTO.0b013e3181ce3e22. PMID 20150827
- [Result] Li XN, Qiu D, Pan X, Hou XX. Mutation of the epidermal growth factor receptor gene and its impact on the efficacy of gefitinib in advanced non-small cell lung cance. Int J Clin Exp Med. 2015 Apr 15;8(4):5397-405. eCollection 2015. PMID 26131116